CLINICAL TRIAL: NCT03531658
Title: Singapore PREconception Study of Long-Term Maternal and Child Outcomes (S-PRESTO)
Brief Title: Singapore PREconception Study of Long-Term Maternal and Child Outcomes
Acronym: S-PRESTO
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University Health System, Singapore (Other); Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Jerry Chan, Prof, KK Women's and Children's Hospital
Other Study IDs: 2019/2143/D; NMRC/TCR/012-NUHS/2014 (Other Grant/Funding Number: National Medical Research Council); MOH-000504 (Other Grant/Funding Number: National Medical Research Council)
Record Dates: First submitted 2017-08-27; First posted 2018-05-22 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Disease; Neurological and Mental Health Conditions; Genetics Predisposition; Skin Condition; Environmental Exposure; Socioeconomic Factors; Psychology, Social
Keywords: Cohort Study; Birth Cohort; Longitudinal Study; Pregnancy; Growth; Developmental Origins of Health and Disease; DOHaD; Epidemiology; Maternal Health; Infant Health; Child Health; Health Outcomes; Postnatal Exposure; Perinatal Exposure; Environmental Factors; Nutrition; Genetics
MeSH Terms: conditions — Metabolic Diseases; Neurologic Manifestations; Genetic Predisposition to Disease; Skin Diseases; Developmental Origins of Health and Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human biological materials such as blood, urine, buccal swabs, saliva, hair, stool, skin microbiome, epithelial swabs (including vaginal, vulval, rectal and breast skin swabs), nasal swabs, breast milk, cord and cord blood, placental samples, subcutaneous fat samples, heel prick blood are collected prospectively from the participants (mother or child) at respective time points, upon their consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
We aim to test the following primary hypothesis that nutrition, lifestyle, and maternal emotional health prior to pregnancy and/or during the first trimester alter the expression of metabolic or neurodevelopmental endophenotypes with accompanying effects on the epigenome/transcriptome of the offspring.

DETAILED DESCRIPTION:
It is now evident that prenatal stage represents a window of susceptibility for early life exposure that can have an effect on developing fetus, with potential long-lasting consequences for offspring growth and development. Emerging research suggest that the environmental modulation of tissue development and function may even occur both before and soon after conception but as yet, limited study has been conducted to investigate the relationship of preconception and early prenatal life conditions, including nutrition, lifestyle and environmental factors, with maternal and offspring health.

This prospective preconception cohort study recruited 1054 women who plan to get pregnant. The investigators will assess the women metabolically, nutritionally and epigenetically, then monitor them from their first missed menses with nutritional surveys and assays and repeated bio-sampling to birth followed by assessment in the women of lactation and lactational nutrition. Biochemical and molecular analyses will be done on the cord and placenta at birth and in buccal smears at frequent postnatal intervals. The women's partners will also be recruited on consent. Phenotypic measures of body composition and core neurodevelopmental measures will be followed in the offspring from birth until 9 years of age. Metabolic and mental health of women will also be measured from preconception until 9 years postpartum. At delivery phase, there are 373 mother-child pairs with 80% of fathers enrolled in the study as well.

This study allows understanding of the potential triggers during early life environment, including nutritional and lifestyle factors, emotional wellbeing, socio-economic status, microbiome, pollutants, metabolomics and epigenetics, which can independently or collectively influence metabolic and neural phenotypes in the offspring and mother. This will help to establish what future directions may hold in terms of possible preventive strategies that may lead to decreased prevalence of metabolic diseases and mental/ neurological disorders.

ELIGIBILITY:
Inclusion Criteria of Mother Participants:

1. Women aged 18-35 years
2. Intention to reside in Singapore for the next 5 years
3. Chinese, Malay, Indian or any combinations of these 3 ethnic groups
4. Planning to conceive within 1 year
5. Able to provide written, informed consent

Exclusion Criteria of Mother Participants:

1. Have been actively trying to conceive for more than 18 months
2. Currently pregnant
3. Assisted fertility, apart from those taking clomiphene alone in the past 1 month
4. Established pre-existing diabetes (type 1 or type 2)
5. Oral or implanted contraception, or with an IUCD in situ in the past 1 month
6. On systemic steroids in the past 1 month
7. On anticonvulsants in the past 1 month
8. On HIV or Hepatitis B or C medication in the past 1 month
9. Not becoming pregnant after more than 12 months from recruitment
10. Eventual multiple pregnancies
11. Pregnancy complications such as miscarriages, ectopic pregnancy, still birth

The partners of the women will also be invited to participate in the study. Babies born from these mothers will be followed up until the child is 9 years of age.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy women aged between 18 and 35 who are actively planning to conceive within a 1-year time frame upon recruitment, and later along with their children born from the indexed pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 1054 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Offspring adiposity | From birth until 9 years of age
  Offspring adiposity (total and percentage fat mass) measured by skinfold calipers, air-displacement plethysmography, quantitative magnetic resonance (QMR), Bioelectrical Impedance Analysis (BIA), and Magnetic resonance imaging (MRI).
Offspring neurocognitive and behavioural development | From 3-12 months up till 9 years of age
  Offspring neurocognitive and behavioural development measured by questionnaires, behavioural tasks and brain MRI.

SECONDARY OUTCOMES:
Duration of gestation | Up to 42 weeks, between estimated date of conception based on ultrasound scan and date of delivery
Fetal growth measured by ultrasound scan | Up to 30 weeks, between 6-36 weeks of gestation
Offspring body weight measured by calibrated weighing scale | From birth until 9 years of age
Offspring pubertal assessment | From 7 until 9 years of age
  Pubertal assessment by Tanner staging
Offspring growth trajectories | From birth until 9 years of age
Offspring adiposity trajectories (total and percentage fat mass) | From birth until 9 years of age
Offspring anogenital distance measured by Vernier calipers | Up to 12 months, from birth until 12 months of age
Offspring allergic wellbeing measured by skin examination and skin prick test | Up to 60 months, from 1 week until 5 years of age
Offspring skin microbiome collected by sterile tape strips | Up to 60 months, from 1 week until 5 years of age
Offspring metabolomics, lipidomics and pollutant profile measured through biospecimens such as cord, cord blood, heel prick blood, and hair samples | From birth until 9 years of age
Offspring epigenetic profile measured through cord, cord blood, and buccal smear samples | From birth until 9 years of age
Offspring gut microbiome measured through stool samples | From birth until 9 years of age
Maternal glucose tolerance status measured by Oral Glucose Tolerance Test (OGTT) | At preconception, 27-28 weeks of gestation, 3 months and 2, 3, 4, 6, 8 years postpartum
Maternal weight measured by calibrated weighing scale | Between preconception, pregnancy and 9 years postpartum
Changes in maternal weight before, during and after gestation | Between preconception, pregnancy and 9 years postpartum
Maternal body weight status determined by body mass index based on weight (kg) /height (m)2 | At preconception visit; 3 months-9 years postpartum
Maternal body composition measured by skinfold calipers, air-displacement plethysmography, bioelectrical impedance analysis and dual-energy X-ray absorptiometry (DXA) | Up to 123 months, between preconception, pregnancy (only using skinfold caliper) and 8 years postpartum
Changes in maternal body composition before, during and after gestation | Up to 123 months, between preconception, pregnancy and 8 years postpartum
Maternal cardiovascular health (subsample) measured through clinical examination | At preconception, 27-28 weeks of gestation, 6 months postpartum
Maternal blood pressure measured by semi-automatic blood pressure device | Between preconception, pregnancy and 9 years postpartum
Maternal allergic wellbeing measured by questionnaires and skin prick test | Up to 40 months, between preconception, pregnancy and 18 months postpartum
Maternal skin microbiome collected by sterile tape strips | 34-36 weeks of gestation and 18 months postpartum
Maternal mental health/emotional wellbeing measured by questionnaires and behavioural tasks | Between preconception, pregnancy and 9 years postpartum
Mode of delivery | Delivery
Pregnancy complications obtained from questionnaires and clinical documents | Up to 41 weeks, between early pregnancy and delivery
Time to pregnancy | Up to 12 months, between the date of last menstrual period obtained from the first preconception visit and before conception (if pregnant) or the most recent follow up (if not pregnant)
Pregnancy and live birth rates based on ultrasound scan | Between early pregnancy and delivery
Maternal metabolomics, lipidomics and pollutant profile measured from biospecimens such as blood, urine, hair | From preconception to pregnancy and up to 8 years postpartum
Maternal epigenetic profile measured from blood and buccal smear samples | From preconception to pregnancy and up to 8 years postpartum
Maternal transcription profile measured from blood samples | From preconception to pregnancy and up to 8 years postpartum
Maternal, paternal and offspring genotyping (blood or buccal samples) | From preconception to pregnancy and up to 8 years postpartum
Maternal micronutrient status measured from blood samples | From preconception to pregnancy and up to 8 years postpartum
Maternal microbiota composition profile measured from stool and epithelial (breast, vaginal and rectal) swab samples | Up to 24 months, preconception, to pregnancy, pre-delivery and 6 weeks postpartum
Breast milk macronutrient profile | Up to 6 months, from 1 week to 6 months postpartum
Breast milk micronutrient profile | Up to 6 months, from 1 week to 6 months postpartum
Breast milk metabolomic profile | Up to 6 months, from 1 week to 6 months postpartum
Breast milk epigenetic profile | Up to 6 months, from 1 week to 6 months postpartum
Maternal and infant transcriptomics (including of breast milk) | Up to 28 months, between preconception, pregnancy and 6 months postpartum
Influence of parental and offspring genotypes, body compositions, lifestyle and diet on the above primary and secondary outcomes | Between preconception, pregnancy and 9 years postpartum

OTHER OUTCOMES:
Offspring health obtained from questionnaires and clinical documents | From birth until 9 years of age
Maternal health obtained from questionnaires and clinical documents | Between preconception, pregnancy and 9 years postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Kok Yen Chan, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loo EXL, Soh SE, Loy SL, Ng S, Tint MT, Chan SY, Huang JY, Yap F, Tan KH, Chern BSM, Tan HH, Meaney MJ, Karnani N, Godfrey KM, Lee YS, Chan JKY, Gluckman PD, Chong YS, Shek LP, Eriksson JG; S-PRESTO Study Group; Chia A, Fogel AM, Goh AEN, Chu AHY, Rifkin-Graboi A, Qiu A, Lee BW, Cheon BK, Vaz C, Henry CJ, Forde CG, Chi C, Koh DXP, Phua DY, Loh DNL, Quah EPL, Tham EH, Law ECN, Magkos F, Mueller-Riemenschneider F, Yeo GSH, Yong HEJ, Chen HY, Tan HH, Pan H, Bever HPSV, Tan HM, Aris IBM, Tay J, Chan JKY, Xu J, Yoong JS, Eriksson JG, Choo JTL, Bernard JY, Huang JY, Lai JS, Tan KML, Godfrey KM, Kwek KYC, McCrickerd K, Narasimhan K, Chong KW, Lee KJ, Chen L, Ling LH, Chen LW, Daniel LM, Shek LP, Fortier MV, Chong MF, Chua MC, Leow MK, Kee MZL, Gong M, Tint MT, Michael N, Lek N, Teoh OH, Mishra P, Li QLJ, Velan SS, Ang SB, Cai S, Goh SH, Lim SB, Tsotsi S, Hsu SC, Toh SES, Sadananthan SA, Tan TH, Yew TW, Gupta V, Rajadurai VS, Han WM, Pang WW, Yuan WL, Zhu Y, Cheung YB, Chan YH, Cheng ZR. Cohort profile: Singapore Preconception Study of Long-Term Maternal and Child Outcomes (S-PRESTO). Eur J Epidemiol. 2021 Jan;36(1):129-142. doi: 10.1007/s10654-020-00697-2. Epub 2020 Nov 21. PMID 33222050
- [Derived] Chu AHY, Padmapriya N, Tan SL, Goh CMJL, Chong YS, Shek LP, Tan KH, Gluckman PD, Yap FKP, Lee YS, Loy SL, Chan JKY, Godfrey KM, Eriksson JG, Chan SY, Bernard JY, Muller-Riemenschneider F. Preconception to postpartum accelerometry-based 24-hour movement behaviors: a prospective cohort study. BMC Public Health. 2026 Jan 7;26(1):465. doi: 10.1186/s12889-025-26034-4. PMID 41501702
- [Derived] Ku CW, Chan HG, Sia AL, Huang C, Quek J, Cheung YB, Tan KML, Lai JS, Godfrey KM, Chan JKY, Yap F, Loy SL. One-carbon metabolism, insulin resistance, and fecundability in a Singapore prospective preconception cohort study. Am J Clin Nutr. 2025 Jul;122(1):335-343. doi: 10.1016/j.ajcnut.2025.04.035. Epub 2025 May 5. PMID 40334751
- [Derived] Chen L, Mir SA, Bendt AK, Chua EWL, Narasimhan K, Tan KM, Loy SL, Tan KH, Shek LP, Chan J, Yap F, Meaney MJ, Chan SY, Chong YS, Gluckman PD, Eriksson JG, Karnani N, Wenk MR. Plasma lipidomic profiling reveals metabolic adaptations to pregnancy and signatures of cardiometabolic risk: a preconception and longitudinal cohort study. BMC Med. 2023 Feb 13;21(1):53. doi: 10.1186/s12916-023-02740-x. PMID 36782297
- [Derived] Li LJ, Du R, Loy SL, Chong YS, Chan JKY, Wong TY, Eriksson JG, Huang Z, Zhang C. Retinal microvasculature and risk of spontaneous abortion in multiethnic Southeast Asian women. Fertil Steril. 2022 Oct;118(4):748-757. doi: 10.1016/j.fertnstert.2022.06.033. Epub 2022 Aug 16. PMID 35981917
- [Derived] Lim SX, Loy SL, Colega MT, Lai JS, Godfrey KM, Lee YS, Tan KH, Yap F, Shek LP, Chong YS, Eriksson JG, Chan JKY, Chan SY, Chong MF. Prepregnancy adherence to plant-based diet indices and exploratory dietary patterns in relation to fecundability. Am J Clin Nutr. 2022 Feb 9;115(2):559-569. doi: 10.1093/ajcn/nqab344. PMID 34626169
- [Derived] Huang L, Loy SL, Chen WQ, Eriksson JG, Chong YS, Huang Z, Chan JKY, Wong TY, Kramer M, Zhang C, Li LJ. Retinal microvasculature and time to pregnancy in a multi-ethnic pre-conception cohort in Singapore. Hum Reprod. 2021 Oct 18;36(11):2935-2947. doi: 10.1093/humrep/deab197. PMID 34492112
- [Derived] Lim SX, Colega MT, M Ayob MN, Robinson SM, Godfrey KM, Bernard JY, Lee YS, Tan KH, Yap F, Shek LP, Chong YS, Eriksson JG, Chan JK, Chan SY, Chong MF. Identification and reproducibility of dietary patterns assessed with a FFQ among women planning pregnancy. Public Health Nutr. 2021 Jun;24(9):2437-2446. doi: 10.1017/S1368980021001178. Epub 2021 Mar 22. PMID 33745499
- [Derived] Loy SL, Ku CW, Lai AEQ, Choo XH, Ho AHM, Cheung YB, Godfrey KM, Chong YS, Gluckman PD, Shek LP, Tan KH, Yap FKP, Chan SY, Chan JKY. Plasma glycemic measures and fecundability in a Singapore preconception cohort study. Fertil Steril. 2021 Jan;115(1):138-147. doi: 10.1016/j.fertnstert.2020.07.014. Epub 2020 Oct 15. PMID 33070964
- See also: Study website — https://www.gusto.sg